CLINICAL TRIAL: NCT07398287
Title: Effect of L-menthol on Breathlessness and Exercise Capacity in Interstitial Lung Disease: a Randomized Crossover Trial
Brief Title: Efficacy of L-menthol on Breathlessness in Interstitial Lung Disease
Acronym: Ment-ILD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Blekinge Institute of Technology (Other); Blekingesjukhuset, Karlskrona (Unknown); Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Ment-ILD
Record Dates: First submitted 2026-01-13; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: interstitial lung disease; breathlessness; dyspnea; CPET; exercise
MeSH Terms: conditions — Lung Diseases, Interstitial; Dyspnea; Motor Activity | interventions — Menthol

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized (ratio 1:1), placebo-controlled, crossover trial (RCT) design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Menthol (Experimental): In the trial, prior to performing submaximal cardio-pulmonary exercise testing (CPET), participants will be administered, L-menthol patch which will be attached to the inside of a facemask that is connected to the breathing circuit.
  Interventions: Drug: L-menthol
- Placebo (Placebo Comparator): For placebo, the patch will contain a similarly patch with strawberry scent.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-menthol — (Sigma-Aldrich, St. Louis, US)
  Arms: L-Menthol
Other: Placebo — Strawberry scent (Sigma-Aldrich, St. Louis, US)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of L-menthol on breathlessness and exercise capacity in patients with Interstitial lung disease (ILD).

DETAILED DESCRIPTION:
Dyspnea is a cardinal symptom in patients with interstitial lung disease (ILD), often triggered by daily-life physical activities. To date, an effective pharmacologic treatment to relieve chronic dyspnea is lacking. Recent pilot data support that inhaled L-menthol can markedly decrease laboratory-induced dyspnea in ILD patients, likely through increased afferent feedback of airflow in the airways by inducing a cooling sensation through olfactory stimulation. The aim of this study is therefore to assess the effectiveness and mechanisms of inhaled menthol for relief of chronic dyspnea in patients with ILD.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study
* Physician diagnosis of fibrosing ILD according to international guidelines
* age 18 years or older
* able to cycle
* able to understand and talk Swedish to participate in the study procedures, as judged by the Investigators.

Exclusion Criteria:

* Resting peripheral oxygen saturation (SpO2) < 92%
* hospitalization or clinical instability during the last four weeks
* treatment with supplementary oxygen at rest or during exercise
* contraindication to exercise testing in accordance with clinical practice guidelines
* expected survival shorter than six months as judged by the Investigator
* medical conditions including congestive heart failure, acute coronary artery disease, neuromuscular diseases, severe psychiatric illness, and olfaction disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Breathlessness intensity | During submaximal test, at isotime during day 2 and day 3.
  The difference between treatment conditions in dyspnea intensity at iso-time. The Borg's modified 0-10 category ratio scale (Borg CR10) will be used, where 0 represents no perceived breathlessness at all, and 10 represents maximum breathlessness intensity ever experienced.

SECONDARY OUTCOMES:
Dyspnea unpleasantness | During submaximal test, at iso-time during day 2 and day 3.
  The difference between treatment conditions in dyspnea unpleasantness at iso-time. The Borg's modified 0-10 category ratio scale (Borg CR10) will be used, where 0 represents no perceived unpleasantness at all, and 10 represents maximum breathlessness unpleasantness ever experienced.
Total time | At the end of submaximal test during day 2 and day 3.
  Time to the limit of tolerance (s) (tLIM)
Exercise capacity | Submaximal test during day 2 and day 3.
  V'O2 (aerobic exercise capacity, absolute and in %pred)
Peak dyspnea intensity | During submaximal test, at peak during day 2 and day 3.
  Dyspnea intensity at peak exercise. The Borg's modified 0-10 category ratio scale (Borg CR10) will be used, where 0 represents no perceived breathlessness at all, and 10 represents maximum breathlessness intensity ever experienced.
Leg fatigue | During submaximal test at day 2 and day 3.
  Leg fatigue. The Borg's modified 0-10 category ratio scale (Borg CR10) will be used, where 0 represents no perceived leg fatigue at all, and 10 represents maximum leg fatigue ever experienced.
Ventilatory efficacy | During submaximal test at day 2 and day 3.
  Efficacy of ventilation (VE/V'CO2-slope)
Saturation | During submaximal test at day 2 and day 3.
  O2-Saturation
Stop reason | During submaximal test at day 2 and day 3.
  Causes of stopping the test
Adverse events | through study completion, an average of 1 week.
  Any adverse events during the test
Respiratory exchange ratio | During the submaximal test at day 2 and day 3.
  Respiratory exchange ratio (RER), defined as V'CO2/V'O2
Heart rate | During the submaximal test at day 2 and day 3.
  Heart rate in beats/min
Breathing frequency | During the submaximal test at day 2 and day 3.
  Breathing frequency in breaths/min
Minute ventilation | During the submaximal test at day 2 and day 3.
  Minute ventilation
Tidal volume (VT) | During the submaximal test at day 2 and day 3.
  Tidal volume in liters
Ventilatory reserve | During the submaximal test at day 2 and day 3.
  defined as maximal voluntary ventilation (MVV) - VE

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Ahmadi, Principal Investigator — Region Skåne and Lund University
Locations (2):
- Sweden (2):
  - Blekinge Institute of Technology, Karlskrona, Blekinge County
  - Lund University hospital and Region Skåne, Lund

IPD SHARING:
Plan to Share IPD: No